CLINICAL TRIAL: NCT03494023
Title: Endoscopic Ultrasound Evaluation of the Common Bile Duct in Patients With Obstructive Jaundice Due to Bilio-Pancreatic Malignancies: A Multicenter Prospective Study
Brief Title: EUS Evaluation of CBD Diameter in Malignant Obstructive Jaundice
Acronym: ECCO
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Collaborators: Catholic University, Italy (Other)
Responsible Party: Principal Investigator, Mihai Rimbas, Assistant Professor, Clinical Hospital Colentina
Other Study IDs: Col-gastro 7
Record Dates: First submitted 2018-03-31; First posted 2018-04-11 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Ampulla of Vater Cancer; Jaundice, Obstructive
MeSH Terms: conditions — Pancreatic Neoplasms; Jaundice, Obstructive | interventions — Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound — Measurement of the common bile duct diameter

SUMMARY:
The main objective of the study is to evaluate the size of the common bile duct (CBD) in a large cohort of patients with jaundice secondary to pancreatic head or distal bile duct malignancy undergoing diagnostic EUS for tissue acquisition or evaluation of resectability and to establish factors associated with a dilation of the CBD greater than 15mm.

DETAILED DESCRIPTION:
Rationale: The size of the common bile duct (CBD) may influence the type of stent used and the type of the procedure performed in cases of EUS-guided biliary drainage. However, no data of the size of the CBD in patients with jaundice presenting with a pancreatic head mass or with a distal cholangiocarcinoma/ carcinoma of the ampulla of Vater are available.

Objectives: To evaluate the size of the CBD in a large cohort of patients with jaundice secondary to pancreatic head or distal bile duct malignancy undergoing diagnostic EUS for tissue acquisition or evaluation of resectability and to establish factors associated with a dilation of the CBD greater than 15mm.

Study design: International prospective observational multicenter trial. Study population: Patients ≥18 years old, referred for EUS-guided tissue sampling or evaluation of resectability of a pancreatic, a distal bile duct lesion or a carcinoma of the ampulla of Vater determining obstructive jaundice.

Intervention: EUS examination Main study parameters/endpoints: measurement of the CBD in patients with an obstructive distal biliary mass. Determine the factors associated with a CBD greater than 15mm Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Measurement of the CBD during EUS examination does not add additional risks to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with jaundice and a pancreatic head mass lesion referred for EUS-guided tissue acquisition or staging
* Patients with jaundice and a distal CBD lesion suggestive of cholangiocarcinoma or a carcinoma of the ampulla of Vater referred for EUS-guided tissue acquisition or staging
* Serum bilirubin level ≥3 mg/dL
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Presence of altered anatomy from previous gastric surgery (Billroth II or Roux-en-Y anastomosis)
* Previously performed sphincterotomy, biliary plastic stent or metal stent placement
* Previous percutaneous drainage of the bile duct
* Pregnancy
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns individuals with jaundice with an indication for EUS examination of a pancreatic head solid lesion, a distal CBD mass, or a carcinoma of the ampulla of Vater who undergo diagnostic EUS-guided tissue acquisition or for evaluation of resectability, discovered at previously performed imaging studies. Only patients with a definitive diagnosis of neoplasia will enter in the final analysis. Eligible individuals will be recruited by endosonographers among the centers of the ECCO study group.
Sampling Method: Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Common bile duct diameter | Enrollment over 6 months
  Measurement by endoscopic ultrasound in patients with malignant obstructive jaundice

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Rimbas, MD, PhD, Principal Investigator — Clinical Hospital Colentina
Locations (1):
- Gastroenterology Department, Clinical Hospital Colentina, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No